CLINICAL TRIAL: NCT06464926
Title: A Prospective Randomized Controlled Trial of Chronic Nausea and Vomiting in Patients With Normal Gastric Emptying Using the Enterra® Therapy System
Brief Title: Chronic Nausea and Vomiting in Patients With Normal Gastric Emptying Using the Enterra® Therapy System (NAVIGATE)
Acronym: NAVIGATE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Enterra Medical, Inc. (Industry)
Collaborators: Bright Research Partners (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ENT-CL-5000
Record Dates: First submitted 2024-06-13; First posted 2024-06-18 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Nausea; Vomiting
Keywords: Chronic; Nausea; Vomiting; Gastric Electrical Stimulation
MeSH Terms: conditions — Nausea; Vomiting; Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Intervention Model Description: Assigned to ON or OFF group. ON group receives active therapy immediately after treatment assignment; OFF group receives active therapy after four months of treatment assignment.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Delegated site personnel will be unblinded to subject treatment assignments to appropriately program their Enterra Therapy System, per study requirements. Unblinded site personnel will be the only role delegated the responsibilities of randomizing subjects to a treatment assignment, performing device interrogations, and completing device programming at study visits according to the randomization assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- ON Group (Experimental): Participants assigned to the ON treatment group will begin with specified device programming values at the randomization visit. Device programming values may be adjusted at follow-up study visits during the blinding period.
  At the conclusion of the 4-month visit, participants will have their devices programmed to individualized therapy as determined by the Investigator. Investigators may adjust programming values at additional follow-up study visits.
  Interventions: Device: Enterra Therapy System
- OFF Group (Experimental): Participants assigned to the OFF treatment group will begin with device programming values set to off at the randomization visit. These settings will continue until the 4-month visit.
  At the conclusion of the 4-month visit, participants will receive specified device programming values. Device programming values may be adjusted at follow-up study visits. At the conclusion of the 8-month visit, participants will have their devices programmed to individualized therapy as determined by the Investigator.
  Interventions: Device: Enterra Therapy System

INTERVENTIONS:
Device: Enterra Therapy System — The Enterra Therapy System is a gastric electrical stimulator system consisting of an implantable pulse generator (Enterra II Model 37800 neurostimulator); two implantable unipolar leads (Enterra Model 4351-35 intramuscular); and device programmer (N'Vision Clinician Programmer Model 8840 with Model 8870 Application Card).
  The programmable neurostimulator operates on a sealed battery and electronic circuitry to provide controlled electrical pulse stimulation through the implanted lead system. A clinician programmer is used to program the neurostimulator and adjust stimulation settings to programmable parameters and stimulation options.

SUMMARY:
The purpose of this research study is to determine if the Enterra® Therapy System can decrease nausea and vomiting symptoms and improve the quality of life for patients with chronic nausea, with or without vomiting, that have normal gastric emptying.

DETAILED DESCRIPTION:
Participants in this study will have an Enterra® Therapy System implanted and be assigned to a study group. Participants will answer daily questions about their nausea and vomiting symptoms and quality of life impacts with their smart device. Participants will answer quality of life questionnaires about their symptoms at study visits. Participants will be involved in this study for approximately twelve months after their study group is assigned.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to complete the informed consent process
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Aged ≥18 years at time of informed consent
* Chronic, drug-refractory nausea that: a) has been present for more than 6 months, and b) has been active within the last 3 months prior to consent
* Patient is able to complete ANMS GCSI-DD surveys on a compatible smart device with: a) a minimum of four (4) ANMS GCSI-DD entries per week for two consecutive weeks, and b) an average ANMS GCSI-DD score for nausea severity of ≥2.5 during the same two-week period
* Refractory or intolerant to two or more of the following antiemetic drug classes: antihistamines, phenothiazines, serotonin type 3 receptor antagonists, dopamine type 2 receptor antagonists, anticholinergics, neurokinin receptor antagonists
* Medically stable, in the opinion of the investigator, during the month prior to consent, with no planned modifications to medical therapy during the course of the study
* Normal gastric emptying as assessed by a qualifying gastric emptying test performed within 2 years of consent if no prior pyloric transection therapy, or within 2 years of consent and after the most recent pyloric transection therapy
* Normal upper endoscopy within 1 year prior to consent (e.g., absence of obstructions, ulcers, or cancers in the esophagus, stomach, or duodenum) performed within 1 year of consent if no prior pyloric transection therapy, or within 1 year of consent and after the most recent pyloric transection therapy

Exclusion Criteria:

* Cognitive impairment or other characteristic that would limit a patient's ability to complete study requirements
* Pyloric transection therapy completed within 1 year of consent
* Documented gastrointestinal (GI) obstruction or pseudo-obstruction
* History of primary swallowing disorders
* History of primary psychogenic vomiting
* History of primary eating disorder
* History of cyclic vomiting syndrome
* History of rumination syndrome
* History of scleroderma
* History of amyloidosis
* History of cannabis hyperemesis syndrome
* Active H. pylori infection
* Evidence of bezoar during most recent endoscopy
* Previous gastric surgery of any type other than a pyloric transection therapy (i.e., pyloroplasty, pyloromyotomy, POP, or G-POEM)
* Uncontrolled thyroid disorder, in the opinion of the investigator
* History of seizures disorders
* Hemoglobin A1c >8.0%
* Peritoneal dialysis or unstable hemodialysis
* Parenteral or enteral nutritional support
* Active pancreatitis
* History of organ transplant, gross malabsorptive syndromes, celiac disease, or inflammatory bowel disease
* Other GI tract diseases and disorders that the investigator believes may have caused the patient's drug-refractory nausea and/or vomiting
* Malignancy (with the exception of basal cell carcinoma of the skin) currently present, initially diagnosed or recurring within 5 years of consent
* Opioid use
* Current cannabis/cannabinoid use that exceeds: 3 days of usage per week, or 2 occurrences during each day of use, or 3 grams of total usage per week
* Heavy alcohol use, defined as: for men, consuming five or more drinks on any day or 15 or more per week; for women, consuming four or more drinks on any day or 8 or more per week
* Injection of Botox into the pyloric sphincter within 6 months of consent
* Active major levels of anxiety/depression, as determined by the investigator
* History of other clinically significant disease, or any other condition which, in the opinion of the Investigator, would jeopardize the safety of the patient or impact the validity of the study results
* Life expectancy <1 year
* Pregnant or breastfeeding at the time of consent or intend to become pregnant during the study
* Any underlying disease leading to follow-up by MRI outside of current MR conditional indications
* Glucagon-like peptide 1 (GLP-1) agonist drug use within 6 months of consent
* Participation in other investigational clinical studies
* Existing or prior gastric electrical stimulator implantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Estimated)
Dates: Start 2025-06-23 (Actual); Primary Completion 2030-06 (Estimated); Study Completion 2030-06 (Estimated)

PRIMARY OUTCOMES:
Change in Nausea Severity Score | 4 Months
  As measured by the American Neurogastroenterology and Motility Society Gastroparesis Cardinal Symptom Index-Daily Diary (ANMS GCSI-DD) nausea severity score

SECONDARY OUTCOMES:
Change in Vomiting Absolute Frequency | 4 Months
  As measured by the American Neurogastroenterology and Motility Society Gastroparesis Cardinal Symptom Index-Daily Diary (ANMS GCSI-DD) weekly vomiting absolute frequency. Analysis only performed if ≥64 evaluable participants have a baseline weekly vomiting frequency of ≥5 per week
Change in Nausea Severity Score | 12 Months
  As measured by the American Neurogastroenterology and Motility Society Gastroparesis Cardinal Symptom Index-Daily Diary (ANMS GCSI-DD) nausea severity score
Change in Vomiting Absolute Frequency | 12 Months
  As measured by the American Neurogastroenterology and Motility Society Gastroparesis Cardinal Symptom Index-Daily Diary (ANMS GCSI-DD) weekly vomiting absolute frequency. Analysis only performed if ≥64 evaluable participants have a baseline weekly vomiting frequency of ≥5 per week
Change in Total Symptom Score | 4 Months
  As measured by the American Neurogastroenterology and Motility Society Gastroparesis Cardinal Symptom Index-Daily Diary (ANMS GCSI-DD) total symptom score
Change in Total Symptom Score | 12 Months
  As measured by the American Neurogastroenterology and Motility Society Gastroparesis Cardinal Symptom Index-Daily Diary (ANMS GCSI-DD) total symptom score
Change in Quality of Life Score | 12 Months
  As measured by the Patient Assessment of Upper Gastrointestinal Disorders Quality of Life (PAGI-QoL) score
Change in Quality of Life Score | 4 Months
  As measured by the Patient Assessment of Upper Gastrointestinal Disorders Quality of Life (PAGI-QoL) score
Change in Early Satiety Score | 4 Months
  As measured by the American Neurogastroenterology and Motility Society Gastroparesis Cardinal Symptom Index-Daily Diary (ANMS GCSI-DD) early satiety score
Change in Postprandial Fullness Score | 4 Months
  As measured by the American Neurogastroenterology and Motility Society Gastroparesis Cardinal Symptom Index-Daily Diary (ANMS GCSI-DD) postprandial fullness score
Change in Abdominal Pain Score | 4 Months
  As measured by the American Neurogastroenterology and Motility Society Gastroparesis Cardinal Symptom Index-Daily Diary (ANMS GCSI-DD) abdominal pain score

CONTACTS AND LOCATIONS:
Overall Officials: Jason Hamann, PhD, Study Director — Enterra Medical, Inc.
Locations (17):
- United States (11):
  - Mayo Clinic Arizona, Scottsdale, Arizona
  - Hoag Hospital, Newport Beach, California
  - Sutter Health, San Francisco, California
  - University of South Florida, Tampa, Florida
  - Endeavor Health, Evanston, Illinois
  - Indiana University Health, Indianapolis, Indiana
  - University of Louisville, Louisville, Kentucky
  - Hackensack Meridian, Neptune City, New Jersey
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Temple Digestive Disease Center, Philadelphia, Pennsylvania
  - Baylor College of Medicine, Houston, Texas
- UZ Leuven, Leuven, Belgium
- France (4):
  - Hôpital Louis-Mourier, Colombes
  - Hôpital Edouard Herriot - CHU de Lyon, Lyon
  - CHU de Bordeaux, Pessac
  - CHU de Rouen, Rouen
- Sahlgrenska Universitetssjukhuset, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No